CLINICAL TRIAL: NCT00403702
Title: Comparison of Two High-Density Silicone Oils in Complicated Rhegmatogenous Retinal Detachment
Brief Title: Comparison High-density Silicone Oils in Retinal Detachment
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APEC-0021
Record Dates: First submitted 2006-11-02; First posted 2006-11-27 (Estimated); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Retinal Detachment
Keywords: Retinal detachment; proliferative vitreoretinopathy; heavier-than-water internal tamponades
MeSH Terms: conditions — Retinal Detachment; Vitreoretinopathy, Proliferative | interventions — oxane HD; densiron

INTERVENTIONS:
Drug: Oxane HD [oil-RMN3-mixture]
Drug: Densiron [(F6H8)

SUMMARY:
The purpose of the study is to compare the safety, intraocular adverse effects and the anatomic and functional outcome with two endotamponade silicone oil after a 3-month in complex inferior retinal re-detachments.

DETAILED DESCRIPTION:
Five to 10% of retinal detachments progressed to proliferative vitreoretinopathy (PVR), the common more cause of surgical failure of retina detachment.

Despite the use of internal tamponades, the treatment of retinal detachments due to a progressed proliferative vitreoretinopathy (PVR) is still a problem. At present, conventional silicone oil, having a lower specific gravity than water, is an excellent tool in advanced PVR retinal detachment especially of the upper circumference.

In the past, to diminish the re-detachments diverse heavier-than-water density endotamponades were investigated by to use in in cases of inferior PVR. However,heavier-than-water density endotamponades have demonstrated adverse short term effects. (Example: silicon dispersion: hypotension and inflammation)

Recently, two new long-term heavier-than-water internal tamponades were introduced: Oxane HD [oil-RMN3-mixture] and Densiron [mixture of 30.5 vol% perfluorohexyloctane (F6H8) with 69.5 vol% polydimethylsiloxane (silicone oil)], showing satisfying anatomical results and good intraocular tolerance.

In the present study, we will compare the anatomical outcome, functional results and intraocular adverse effects of two types of heavier tamponades.

ELIGIBILITY:
Inclusion Criteria:

* Patients complicated persistent retinal detachment due secondary to proliferative vitreoretinopathy

Exclusion Criteria:

* Diabetes
* Uveitis
* Glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-08 (Actual); Primary Completion 2006-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
visual acuity
anatomical results

SECONDARY OUTCOMES:
complication: hypotony,
vitreous hemorrhage,
inflammatory reaction,
cataract,
chronic hypotony,
IOP elevated intraocular pressure,
pseudohypopyon,
fibrin,
emulsification droplets in the anterior chamber

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Quiroz-Mercado, MD, Study Director — Asociación para Evitar la Ceguera en México
Locations (1):
- Asociacion Para Evitar la Ceguera en Mexico, México, D.F, Mexico

REFERENCES:
- [Background] Sandner D, Engelmann K. First experiences with high-density silicone oil (Densiron) as an intraocular tamponade in complex retinal detachment. Graefes Arch Clin Exp Ophthalmol. 2006 May;244(5):609-19. doi: 10.1007/s00417-005-0110-8. Epub 2005 Oct 5. PMID 16205937
- [Background] Theelen T, Tilanus MA, Klevering BJ. Intraocular inflammation following endotamponade with high-density silicone oil. Graefes Arch Clin Exp Ophthalmol. 2004 Jul;242(7):617-20. doi: 10.1007/s00417-004-0898-7. Epub 2004 Mar 17. PMID 15029505
- [Background] Nicolai U, Eckardt C, Kohlhoff M, Wottge HU. Biocompatibility of silicone oil and high-density liquids. An immunologic study. Ger J Ophthalmol. 1992;1(3-4):180-7. PMID 1483133
- [Background] Mester U, Rothe R, Zubcov A. Experimental studies with a high-density silicone oil for giant retinal tear. Ophthalmic Res. 1986;18(2):81-6. doi: 10.1159/000265419. PMID 3737116
- [Background] Wong D, Cazabon S, Ali H, Kumar I, Valldeperas X, Groenewald C, Pearce I. Can the sequential use of conventional silicone oil and heavy oil be a strategy for the management of proliferative vitreoretinopathy? Ann Acad Med Singap. 2006 Mar;35(3):181-4. PMID 16625267
- [Background] Scheer S, Boni S, Barale PO, Bourhis A, Bonnel S, Tuil E, Girmens JF, Buil O, Baudouin C, Laroche L, Nordmann JP, Poisson F, Warnet JM, Sahel JA. [Heavy silicone oil as internal tamponade for retinal detachment: efficacy and tolerance]. J Fr Ophtalmol. 2006 Feb;29(2):129-35. doi: 10.1016/s0181-5512(06)73760-3. French. PMID 16523153
- [Background] Tognetto D, Minutola D, Sanguinetti G, Ravalico G. Anatomical and functional outcomes after heavy silicone oil tamponade in vitreoretinal surgery for complicated retinal detachment: a pilot study. Ophthalmology. 2005 Sep;112(9):1574. doi: 10.1016/j.ophtha.2005.04.013. PMID 16139666
- [Background] Bhisitkul RB, Gonzalez VH. "Heavy oil" for intraocular tamponade in retinal detachment surgery. Br J Ophthalmol. 2005 Jun;89(6):649-50. doi: 10.1136/bjo.2004.057182. No abstract available. PMID 15923493
- [Background] Wolf S, Schon V, Meier P, Wiedemann P. Silicone oil-RMN3 mixture ("heavy silicone oil") as internal tamponade for complicated retinal detachment. Retina. 2003 Jun;23(3):335-42. doi: 10.1097/00006982-200306000-00008. PMID 12824833
- [Background] Rizzo S, Genovesi-Ebert F, Belting C, Vento A, Cresti F. A pilot study on the use of silicone oil-RMN3 as heavier-than-water endotamponade agent. Graefes Arch Clin Exp Ophthalmol. 2005 Nov;243(11):1153-7. doi: 10.1007/s00417-005-0015-6. Epub 2005 Jun 28. PMID 15983817
- [Derived] Schwartz SG, Flynn HW Jr, Wang X, Kuriyan AE, Abariga SA, Lee WH. Tamponade in surgery for retinal detachment associated with proliferative vitreoretinopathy. Cochrane Database Syst Rev. 2020 May 13;5(5):CD006126. doi: 10.1002/14651858.CD006126.pub4. PMID 32408387